CLINICAL TRIAL: NCT06213896
Title: Screening And Detecting Eye Diseases With Hybrid Deep Learning Algorithms From Fundus Images And Validation Of Automated Artificial Intelligence Algorithm
Brief Title: Detecting Eye Diseases Via Hybrid Deep Learning Algorithms From Fundus Images
Status: Completed | Type: Observational
Sponsor: Ural Telekomunikasyon Sanayi Ticaret Anonim Sirketi (Industry)
Responsible Party: Sponsor
Other Study IDs: EC-2023-TR
Record Dates: First submitted 2024-01-09; First posted 2024-01-19 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-01

CONDITIONS: Glaucoma; Age-Related Macular Degeneration; Retinal Vein Occlusion; Diabetic Retinopathy; Diabetic Macular Edema; Eye Diseases
Keywords: Artificial Intelligence; Eye Diseases
MeSH Terms: conditions — Glaucoma; Macular Degeneration; Retinal Vein Occlusion; Diabetic Retinopathy; Eye Diseases | interventions — Mydriatics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Mydriatic Agent — Subjects will be administered mydriatic medication to dilate their pupils.
  Other Names: Tropicamide drops
Procedure: Color Fundus Photography — Subjects will undergo fundus photography before and after administration of mydriatic agent.
Device: EyeCheckup v2.0 — Screening for existence of eye diseases

SUMMARY:
Eye health is of great importance for quality of life. Some eye diseases can progress and cause permanent damage up to vision loss if they are not treated early. Therefore, it is of great importance to have regular eye examinations and to detect possible eye diseases before they progress. Healthy people should also undergo eye screening once a year, and those with any complaints regarding eye health should be examined.

With the advancing technology, Artificial Intelligence (AI) has begun to play a significant role in the healthcare sector. Retinal diseases, serious health problems resulting from damage to the back part of the eye's retina, include conditions such as retinopathy, macular degeneration, and glaucoma. Artificial intelligence, with its visual recognition and analysis capabilities, holds great potential in the early diagnosis of retinal diseases.

AI-based diagnosis of retinal diseases typically involves the use of specialized algorithms that analyze retinal images. These algorithms identify abnormal features in the eye, providing doctors with a quick and accurate diagnosis.

EyeCheckup v2.0 will diagnose glaucoma suspicion, severe glaucoma suspicion, age-related macular degeneration diagnosis, RVO diagnosis, diabetic retinopathy diagnosis and stage, presence/absence of DME suspicion and other retinal diseases from fundus images. This study is designed to assess the safety and efficacy of EyeCheckup v2.0.

The study is a single center study to determine the sensitivity and specificity of EyeCheckup to retinal and optic disc diseases. EyeCheckup v2.0 is an automated software device that is designed to analyze ocular fundus digital color photographs taken in frontline primary care settings in order to quickly screen.

DETAILED DESCRIPTION:
According to the World Health Organization's worldwide report published in 2020, at least 2.2 billion people worldwide currently have visual impairment, and at least 1 billion of them have a visual impairment that can be prevented or has not yet been addressed. The world faces significant eye health challenges, including inequalities in the coverage and quality of eye care prevention, treatment, and rehabilitation services, a lack of trained eye care providers, and poor integration of eye care services into health systems, among others.

It is known that more than 80% of all visual disorders can be prevented or treated. An eye fundus examination must be performed by a retina specialist to make a correct diagnosis, but people only consult an ophthalmologist when they feel any discomfort. While typically symptoms progress so much that once a disease occurs, resulting in expensive treatments and surgeries, often the damage is irreversible, resulting in visual impairment or even permanent vision loss.

Artificial intelligence is used to study and develop theories and methods that can help simulate and extend human intelligence, which have been used in many fields of research such as automatic diagnosis and medicine. In recent years, the intersection of artificial intelligence (AI) technology and modern medicine has made effective and rapid disease screening possible. EyeCheckup is an automated software device designed to analyze digital color photographs of the ocular fundus to quickly screen for retinal and optic disc diseases.

The main aim of the research is to evaluate the performance of the automatic screening algorithm to detect steerable retinal and optic disc diseases based on color fundus images and to determine its sensitivity and specificity towards possible diseases. For the clinical validation of the system, the images will be evaluated by ophthalmologists and the results will be compared with the artificial intelligence algorithm.

After exclusions, this study will enroll up to 1528 subjects that meet the eligibility criteria. Participants who meet the eligibility criteria will be recruited after obtaining written informed consent from primary health care providers. Subjects will undergo fundus photography per, Food and Drug Administration (FDA) cleared, ophthalmic cameras. Images will be taken according to a specific EyeCheckup imaging protocol provided to the ophthalmic camera operator and then analyzed by the EyeCheckup v2.0 device.

Methods and tools to be used in the research:

I. Fundus photo capturing with non-mydriatic cameras: Optic disc-centered and fovea-centered fundus images will be taken with Canon CR-2 AF, Topcon TRC-NW400 and Optomed Aurora Non-mydriatic fundus cameras. For volunteers whose non-mydriatic images cannot be obtained, pupil dilation will be achieved by instilling tropicamide drops, and then images will be taken. Canon CR-2 AF, Topcon TRC-NW400 and Optomed Aurora Non-mydriatic fundus cameras, from which retina images will be taken, are CE marked and FDA approved.

Tests to be done:

I. Fundus images obtained with three different cameras from each volunteer included in the study will be analyzed separately for both the right eye and the left eye by the EyeCheckup artificial intelligence algorithm on a camera-based basis.

ii. Evaluation of Canon CR-2 AF images by retina and glaucoma specialists for clinical validation of the system and comparison of the results,

ELIGIBILITY:
Inclusion Criteria:

Must understand the study and sign informed consent. No history of retinal vascular disease, cataracts or any other disease that may affect the appearance of the retina or optic disc (refractive error and ocular surface disease are allowed).

No history of intraocular surgery or ocular laser treatment for any retinal disease, other than cataract surgery.

18 years and over

Exclusion Criteria:

Not understand the study or informed consent, Media opacity or other defect that would prevent taking a fundus photograph with the feature to be evaluated (which could not be taken with a non-mydriatic fundus camera in 6 attempts or was rejected 6 times by the EyeCheckup quality algorithm due to quality), Has intraocular surgery other than cataracts or has had laser treatment on the retina, Contraindicated for imaging with the fundus imaging systems used in the study, Under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinic invitation to volunteer, Eighteen years of age or older Have been referred to an ophthalmologist for eye examination to screen for eye disease
Sampling Method: Non-Probability Sample
Enrollment: 1528 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-04-18 (Actual)

PRIMARY OUTCOMES:
To determine the accuracy of diagnosis with artificial intelligence algorithm | through study completion, an average of 1 year
  Comparison of the compatibility of the diagnosis of the artificial intelligence algorithm with the diagnoses of retina and glaucoma specialists

SECONDARY OUTCOMES:
To determine the sensitivity and specificity of EyeCheckup v2.0 to detect retinal and optic disc diseases | through study completion, an average of 1 year
  1. To determine the sensitivity of EyeCheckup v2.0 to detect Glaucoma, RVO, diabetic retinopathy, suspected DME, ARMD, other retinal disease (True positive rate of the algorithm)
  2. To determine the specificity of EyeCheckup v2.0 to detect Glaucoma, RVO, diabetic retinopathy, suspected DME, ARMD, other retinal disease (True negative rate of the algorithm)
  3. To determine the specificity of EyeCheckup v2.0 to detect Refere/Nonrefere (True negative rate of the algorithm)
  4. To determine the sensitivity of EyeCheckup v2.0 to detect Refere/Nonrefere (True positive rate of the algorithm)

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University Hospital, Antalya, Turkey (Türkiye)